CLINICAL TRIAL: NCT04435977
Title: Efficacy and Safety of Cabozantinib in Patients With Hepatocellular Carcinoma Progressing on or Intolerant to Prior Treatment With Immune Checkpoint Inhibitors: A Phase II Study (Immunocabo)
Brief Title: Efficacy and Safety of Cabozantinib in Patients With Hepatocellular Carcinoma
Acronym: Immunocabo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2019-002
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Hepatocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: Single group assignement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): Drug: Cabozantinib Subjects who meet all study eligibility criteria will take tablets containing 60 mg of cabozantinib once daily orally. Required dose reductions will be in decrements of 20 mg cabozantinib (maximum two dose reductions).
  Interventions: Drug: Cabozantinib 60 MG

INTERVENTIONS:
Drug: Cabozantinib 60 MG — • The assigned dose for study treatment is 60 mg qd. Two dose reductions will be permitted (Table 2):
  * 60 mg qd to 40 mg qd (level 1)
  * 40 mg qd to 20 mg qd (level 2)

SUMMARY:
This is an open-label, single-center, Phase II trial designed to estimate in terms of PFS the efficacy of cabozantinib, given as second- or third- line treatment in HCC patients that progress on or are intolerant to immune checkpoint inhibitors, including anti-PD-1 and anti-PD-L1 antibodies.

DETAILED DESCRIPTION:
Subjects who meet all study eligibility criteria will take tablets containing 60 mg of cabozantinib once daily orally. Required dose reductions will be in decrements of 20 mg cabozantinib (maximum two dose reductions).

Subjects will receive study treatment as long as they continue to experience clinical benefit in the opinion of the investigator or until there is unacceptable toxicity.

Primary objective of this study is to evaluate the efficacy of cabozantinib, given as second- or third-line treatment in HCC patients that progress on or are intolerant to immune checkpoint inhibitors.

Secondary objectives for this study are as follows:

* To evaluate the activity of cabozantinib, in terms of ORR (CR+PR) as per RECIST 1.1, duration of response, time to treatment failure (TTF), time to progression (TTP), and OS
* To evaluate the safety and tolerability of cabozantinib

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of HCC (results of a previous biopsy will be accepted)
* A baseline tumor tissue (newly obtained) available at screening is optional. Patient must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy according to the treating institution's guidelines and requirements for such procedure. Biopsy cannot be performed less than ten days before treatment start.
* The subject has disease that is not amenable to a locoregional treatment approach (eg, transplant, surgery, radiofrequency ablation, TACE)
* Patients must have documented disease progression following at least 1 and no more than 2 prior systemic regimens for advanced disease (nonresectable or metastatic), the last of which includes immune checkpoint inhibitors. Alternatively, eligible patients may have experienced an immune-related, requiring treatment discontinuation.
* Recovery to ≤ Grade 1 from toxicities related to any prior treatments, unless the adverse events are clinically not significant and/or stable on supportive therapy
* Age ≥ 18 years old on the day of consent
* ECOG performance status of 0 or 1 (See Appendix V)
* Adequate hematologic function, based upon meeting the following laboratory criteria within 7 days before treatment beginning:

  * a. absolute neutrophil count (ANC) ≥ 1200/mm3 (≥ 1.2 x 109/L)
  * b. platelets ≥ 60,000/mm3 (≥ 60 x 109/L)
  * c. hemoglobin ≥ 8 g/dL (≥ 80 g/L)
* Adequate renal function, based upon meeting the following laboratory criteria: serum creatinine ≤ 1.5 × upper limit of normal or calculated creatinine clearance ≥ 40 mL/min (using the Cockroft-Gault equation: (140 - age) x weight (kg)/(serum creatinine × 72 [mg/dL]) for males. (For females multiply by 0.85)
* Child-Pugh Score of A (See Appendix IV)
* Total bilirubin ≤ 2 mg/dL within 7 days before treatment start
* Serum albumin ≥ 2.8 g/dL (≥ 28 g/L) within 7 days before treatment start
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5.0 upper limit of normal (ULN)
* Antiviral therapy per local standard of care if active hepatitis B (HBV) infection
* Capable of understanding and complying with the protocol requirements and signed informed consent
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment
* Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression, low body weight, or other reasons

Exclusion Criteria:

* Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma
* Child-Pugh score of B or C
* Any type of anticancer agent (including investigational) within 2 weeks before treatment start
* Radiation therapy within 4 weeks (2 weeks for radiation for bone metastases) or radionuclide treatment (eg, I-131 or Y-90) within 6 weeks of treatment start. Subject is excluded if there are any clinically relevant ongoing complications from prior radiation therapy
* Prior cabozantinib treatment
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before treatment start. Eligible subjects must be without corticosteroid treatment at the time of treatment start
* Concomitant anticoagulation, at therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, low molecular weight heparin (LMWH), thrombin or coagulation factor X (FXa) inhibitors, or antiplatelet agents (eg, clopidogrel). Low-dose aspirin for cardioprotection (per local applicable guidelines), low-dose warfarin (≤ 1 mg/day), and low-dose LMWH are permitted
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:
* a. Cardiovascular disorders including:

  * i. Symptomatic congestive heart failure, unstable angina pectoris, or serious cardiac arrhythmias
  * ii. Uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic, or > 100 mm Hg diastolic despite optimal antihypertensive treatment
  * iii. Stroke (including TIA), myocardial infarction, or other ischemic event within 6 months before treatment start.
* iv. Thromboembolic event within 3 months before treatment start. Subjects with thromboses of portal/hepatic vasculature attributed to underlying liver disease and/or liver tumor are eligible
* b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

  * i. Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
  * ii. Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before treatment start
  * Note: Complete healing of an intra-abdominal abscess must be confirmed prior to treatment start
* c. Major surgery within 2 months before treatment start. Complete healing from major surgery must have occurred 1 month before treatment start. Complete healing from minor surgery (eg, simple excision, tooth extraction) must have occurred at least 7 days before treatment start. Subjects with clinically relevant complications from prior surgery are not eligible
* d. Cavitating pulmonary lesion(s) or endobronchial disease
* e. Lesion invading a major blood vessel including, but not limited to: inferior vena cava, pulmonary artery, or aorta. Subjects with lesions invading the portal vasculature are eligible
* f. Clinically significant bleeding risk including the following within 3 months of treatment start: hematuria, hematemesis, hemoptysis of >0.5 teaspoon (>2.5 mL) of red blood, or other signs indicative of pulmonary hemorrhage, or history of other significant bleeding if not due to reversible external factors
* g. Other clinically significant disorders such as:

  * i. Active infection requiring systemic treatment, known infection with human immunodeficiency virus (HIV), or known acquired immunodeficiency syndrome (AIDS)-related illness. Subjects with active hepatitis virus infection controlled with antiviral therapy are eligible
  * ii. Serious non-healing wound/ulcer/bone fracture
  * iii. Malabsorption syndrome
  * iv. Uncompensated/symptomatic hypothyroidism
  * v. Requirement for hemodialysis or peritoneal dialysis
  * vi. History of solid organ transplantation
  * vii. Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Subjects with untreated or incompletely treated varices with bleeding or high risk for bleeding. Subjects treated with adequate endoscopic therapy (according to institutional standards)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
PFS | through study completion, an average of 1 year
  PFS on cabozantinib treatment (considering as PFS events: clinical or radiological progressive disease, per RECIST 1.1, or death).

SECONDARY OUTCOMES:
ORR | through study completion, an average of 1 year
  ORR as per RECIST 1.1, duration of response, TTF, TTP, and OS.
safety and tolerability | through study completion, an average of 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Lorenza Rimassa, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No